CLINICAL TRIAL: NCT05031819
Title: Managing Hypertension Among People Living With HIV: An Integrated Model (MAP-IT)
Brief Title: Managing Hypertension Among People Living With HIV
Acronym: MAP-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Dike Ojji (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Dr. Dike Ojji, Professor, University of Abuja
Organization: University of Abuja (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UATH/HREC/PR/2020-009; UH3HL154498 (NIH)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure; Human Immunodeficiency Virus I Infection; Acquired Immunodeficiency Syndrome; Hypertension
Keywords: Noncommunicable Diseases; Cardiovascular Diseases; Health Services Accessibility; HIV; Nigeria
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hypertension; Noncommunicable Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Step wedge design. One group with a cross over.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practice Facilitation to support TASSH integration (group A). (Experimental): Components of the PF strategy include: (a) establishment of a steering committee of key stakeholders (ministry of health, state primary care agency, AIDS control agency, patient advocates) to provide leadership and guide integration of TASSH into HIV care platform; (b) training of the HIV nurses on TASSH protocol; and (c) training of practice facilitators, who will serve as coaches, provide support, and performance feedback to the PHC nurses on TASSH implementation.
  Interventions: Other: Nurse-led Task-Shifting Strategy for Hypertension Control (TASSH) plus Practice Facilitation.
- TASSH only (group B) (Sham Comparator): HIV nurses based at Group B facilities will be trained on the 5As counseling approach strategy (Ask, Assess, Advise, Assist, and Arrange) and referral for the participants to the health center. However, they will not receive practice facilitation from the POFs. Participants attending PHC randomized to Group B will receive standard care offered by the facility.
  Interventions: Other: Nurse-led Task-Shifting Strategy for Hypertension Control (TASSH) plus Practice Facilitation.

INTERVENTIONS:
Other: Nurse-led Task-Shifting Strategy for Hypertension Control (TASSH) plus Practice Facilitation. — * TASSH includes CVD risk assessment; medication initiation and titration; lifestyle counseling and patient referral to physician care for complex cases.
  * Practice Facilitation includes the training of external experts to support the HIV nurses implementing TASSH

SUMMARY:
The Managing Hypertension Among People Living with HIV: An InTegrated Model (MAP-IT) a stepped wedge, cluster-randomized controlled trial to evaluate the effect of practice facilitation (PF) on the integration of a Task-Shifting Strategy for hypertension (HTN) control (TASSH) into HIV care for management of HTN in people living with HIV (PLWH). The study will recruit 960 PLWH across 30 primary health centers (PHCs) in Akwa Ibom State (32 patients/PHC).

DETAILED DESCRIPTION:
People Living with HIV (PLWH) are at increased risk for non-communicable diseases (NCDs) including cardiovascular diseases (CVD) with hypertension (HTN) the most common. Integrating NCD management into HIV chronic care services may be a cost-effective strategy to mitigate the rising burden of NCDs in PLWH. The goal of the study is to evaluate the effectiveness of practice facilitation in the integration of a task-shifting strategy for hypertension control into HIV care service delivered in primary health centers in Akwa Ibom State, Nigeria.

This study will occur in two phases: 1) The first phase is a UG3 Planning Phase during which investigators will use the iPARiHS implementation science framework to explore factors and support systems required for successful implementation and integration of TASSH into existing HIV chronic care platform and development of a context-specific practice facilitation strategy. 2) The second phase, which is the focus of this record, is a UH3 Implementation Phase during which we will use a stepped-wedge, cluster RCT, guided by the RE-AIM implementation science framework, to evaluate the effect of practice facilitation strategy on the level of adoption of TASSH, hypertension control, and level of sustainment of TASSH in management of hypertension among 960 patients enrolled in HIV treatment services across 30 PHCs.

ELIGIBILITY:
Inclusion Criteria:

1. Persons aged 18 years or older
2. Be HIV positive and currently enrolled in HIV treatment services at one of the 30 study PHCs, be receiving HTN treatment services at one of the 30 study PHCs, or can be enrolled at one of the 30 study PHCs to receive HTN services for the entire study duration.
3. Have elevated blood pressure between 140-179 mm Hg systolic and/or 90-109 mm Hg diastolic, as determined by the average of the latter two of three separate BP readings during one clinic visit
4. Able to provide consent

Exclusion Criteria:

1. BP ≥180/100 mm Hg
2. Known history of kidney disease, heart disease, diabetes mellitus, stroke
3. A female who is pregnant or breastfeeding at the time of enrollment
4. Inability to provide informed consent
5. Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
The effect of practice facilitation on the rate of adoption of a task sharing and strengthening strategy (TASSH). | 12 months
  TASSH is defined as: i identification of patients with uncontrolled hypertension; ii measurement of blood pressure and anthropometrics; iii initiation of lifestyle counselling and blood pressure medications; iv. referral of complicated patients

SECONDARY OUTCOMES:
Level of adoption and implementation fidelity of task sharing and strengthening for hypertension. | 12 months
  We will evaluate the level of adoption and implementation fidelity of TASSH as potential mechanisms that may explain the effect of PF on our primary outcome of BP control and change in systolic BP (SBP) from baseline to 12 months.
Level of sustainment of TASSH | 6 months
  We will evaluate the level of sustainment of TASSH at the end of the 6-month follow- up period.

CONTACTS AND LOCATIONS:
Overall Officials: Dike Ojji, MBBS, Ph.D, Principal Investigator — University of Abuja; Olugbenga Ogedegbe, MD, MPH, Principal Investigator — NYU Langone Health; Juliet Iwelunmor, Ph.D, Principal Investigator — St. Louis University; Angela Attah, MBBS, MPH, Principal Investigator — FHI 360; DANIEL HENRY, Study Director — Cardiovascular Research Unit, University of Abuja
Locations (1):
- Primary Health Care Facilities, Uyo, Akwa Ibom State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aifah AA, Hade EM, Colvin C, Henry D, Mishra S, Rakhra A, Onakomaiya D, Ekanem A, Shedul G, Bansal GP, Lew D, Kanneh N, Osagie S, Udoh E, Okon E, Iwelunmor J, Attah A, Ogedegbe G, Ojji D. Study design and protocol of a stepped wedge cluster randomized trial using a practical implementation strategy as a model for hypertension-HIV integration - the MAP-IT trial. Implement Sci. 2023 May 10;18(1):14. doi: 10.1186/s13012-023-01272-5. PMID 37165382
- [Derived] Iwelunmor J, Ogedegbe G, Dulli L, Aifah A, Nwaozuru U, Obiezu-Umeh C, Onakomaiya D, Rakhra A, Mishra S, Colvin CL, Adeoti E, Badejo O, Murray K, Uguru H, Shedul G, Hade EM, Henry D, Igbong A, Lew D, Bansal GP, Ojji D. Organizational readiness to implement task-strengthening strategy for hypertension management among people living with HIV in Nigeria. Implement Sci Commun. 2023 May 4;4(1):47. doi: 10.1186/s43058-023-00425-3. PMID 37143131